CLINICAL TRIAL: NCT06199817
Title: The Effect Of Multiple Occupational Therapies On Functional Remission And Subjective Recovery For Patients With Schizophrenia: A Randomized Controlled Trial
Brief Title: The Effect Of Multiple Occupational Therapies On Functional Remission And Subjective Recovery For Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Merve Uğuryol Ünal, Research Assistant, Phd, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 16-5.1/7
Record Dates: First submitted 2023-12-14; First posted 2024-01-10 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2023-12

CONDITIONS: Occupational Therapy; Schizophrenia; Remission; Well-Being, Psychological
Keywords: Shizophrenic Disorder; Occupational Therapy; Remission; Well-Being, Psychological
MeSH Terms: conditions — Schizophrenia; Psychological Well-Being | interventions — Occupational Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention group was informed about the research. The intervention group consists of patients diagnosed with schizophrenic disorder. Music, sports and garden-soil activities were applied to the intervention group.
  Interventions: Behavioral: occupational therapies
- Control Group (No Intervention): The control group was informed about the research.

INTERVENTIONS:
Behavioral: occupational therapies — music, garden-soil and sports practices for individuals diagnosed with schizophrenic disorder
  Arms: Intervention Group

SUMMARY:
Objective: This study aimed to evaluate the effect of multiple occupational therapies on functional remission and subjective recovery of individuals with schizophrenic disorder. Methods: 26 people with schizophrenic disorder were divided into two groups using a random number table. The intervention group participated in routine community mental health center services and a total of 24 sessions of occupational therapies three times a week, while the control group participated in routine community mental health center services.

DETAILED DESCRIPTION:
Background: Occupational therapies are one of the psycho-social intervention methods used in the treatment of serious mental disorders characterized by disability, such as schizophrenia.

Objective: This study aimed to evaluate the effect of multiple occupational therapies on functional remission and subjective recovery of individuals with schizophrenic disorder.

Methods: 26 people with schizophrenic disorder were divided into two groups using a random number table. The intervention group participated in routine community mental health center services and a total of 24 sessions of occupational therapies three times a week, while the control group participated in routine community mental health center services. Data were collected using the Subjective Recovery Assessment Scale and the Functional Remission of General Schizophrenia Scale.

ELIGIBILITY:
Inclusion Criteria:

* Being in the 18-65 age group
* have been diagnosed with schizophrenia for at least one year
* be in remission of the disease
* volunteering to participate in research
* not have any physical health problems that would prevent their participation in the research

Exclusion Criteria:

* have a physical health problem that prevents participation in the research
* Having a communication problem
* not willing to participate in research

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-08-19 (Actual)

PRIMARY OUTCOMES:
Functional Remission of General Schzophrenia Scale (Pre Test) | 2 month
  The scale is a 5-point Likert type scale consisting of 19 items. The minimum score obtained from the scale is 19 points and the maximum score is 95 points. High scores from the scale indicate high functionality, while low scores from the scale indicate low functionality. Scale scores were expected to be low in the pretest.
Subjective Recovery Assessment Scale (Pre Test) | 2 month
  The scale is a 5-point Likert type consisting of 17 items. The lowest score from the scale is 17 and the highest score is 85. Higher scores from the scale indicate that the individual perceives himself as more improved. Scale scores were expected to be low in the pretest.

SECONDARY OUTCOMES:
Functional Remission of General Schzophrenia Scale (Post Test) | Forth month
  The scale is a 5-point Likert type scale consisting of 19 items. The minimum score obtained from the scale is 19 points and the maximum score is 95 points. High scores from the scale indicate high functionality, while low scores from the scale indicate low functionality. "Functional Remission of General Schzophrenia Scale" score was expected to increase in the post test.
Subjective Recovery Assessment Scale (Post Test) | Forth month
  The scale is a 5-point Likert type consisting of 17 items. The lowest score from the scale is 17 and the highest score is 85. Higher scores from the scale indicate that the individual perceives himself as more improved. It was expected that the score obtained from the scale in the post-test would be high.

OTHER OUTCOMES:
Functional Remission of General Schzophrenia Scale (Follow Up Test) | Seventh month
  The scale is a 5-point Likert type scale consisting of 19 items. The minimum score obtained from the scale is 19 points and the maximum score is 95 points. High scores from the scale indicate high functionality, while low scores from the scale indicate low functionality. "Functional Remission of General Schzophrenia Scale" score was expected to increase in the follow up test.
Subjective Recovery Assessment Scale (Follow Up Test) | Seventh month
  The scale is a 5-point Likert type consisting of 17 items. The lowest score from the scale is 17 and the highest score is 85. Higher scores from the scale indicate that the individual perceives himself as more improved. It was expected that the score obtained from the scale in the follow-up test would be high.
Effect Size of Functional Remission of General Schzophrenia Scale | Seventh month
  It shows how the applied occupational therapies affect the final and follow-up test scale scores of the intervention and control groups in terms of time.
Effect Size of Subjective Recovery Assessment Scale | Seventh month
  It shows how the applied occupational therapies affect the final and follow-up test scale scores of the intervention and control groups in terms of time.

CONTACTS AND LOCATIONS:
Overall Officials: Aysegul Donmez, Study Director — Ege University

IPD SHARING:
Plan to Share IPD: No